CLINICAL TRIAL: NCT06669780
Title: Single-Blind, Randomized, Controlled Pilot Trial of a Cognitive-Behavioral Therapy Digital Therapeutic Delivered Online for Post-Traumatic Headaches in Adults With History of Concussive Traumatic Brain Injury
Brief Title: e-CBT DTx for Post Traumatic Headaches in Adults With History of TBI
Acronym: AMMO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMMO-TBI-2023
Record Dates: First submitted 2024-06-24; First posted 2024-11-01 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-01

CONDITIONS: Post-Traumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active (Experimental): This arm will receive access to an online program that will guide them through cognitive behavioral therapy program.
  Interventions: Device: AMMO PTH DTx
- Sham comparator (Sham Comparator): Participants will obtain access to an online program with activities not including the cognitive behavioral therapy
  Interventions: Device: AMMO SHAM

INTERVENTIONS:
Device: AMMO PTH DTx — An online cognitive behavioral therapy program accessed through a online program.
  Arms: Active
Device: AMMO SHAM — Online activities not including CBT in the AMMO online program.
  Arms: Sham comparator

SUMMARY:
The AMMO digital therapeutic (DTx) study will provide an online based program for participants with migraines after head injury to follow for 12 weeks. This study aims to see if using cognitive behavioral therapy aimed at military service members in an online self administered platform is effective therapy in the relief of migraines compared. The study will use a single blind online comparative program to test the effect.

DETAILED DESCRIPTION:
The AMMO digital therapeutic (DTx) will be a novel intervention for PTH following concussive TBI, therefore this project is a pilot trial designed to test this new treatment. This pilot is a single-blind, randomized, controlled, interventional trial of current and former military personnel along with civilians with a history of concussive TBI and current PTH. The pilot trial will be conducted via online portal accessible by smartphone, tablet, or computer with remote interaction between participants and study staff. The pilot trial will include up to 100 participants randomized to either the active intervention or a comparison condition at a 1:1 ratio, and will provide preliminary data to determine the sample size of a future full clinical trial. Participants will complete a 12 week intervention period followed by a follow-up assessment 4 weeks after intervention is complete. Participants randomized to the comparison group will be provided access to the open label after end of 16 week follow-up.

In addition, updates to the DTx to improve usability and acceptability will be made if necessary based on feedback from the pilot trial, then applied to the final DTx used in a future, larger, clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Be aged ≥ 18 to ≤ 70 years
* Have a history of concussive TBI ≥ 3 months prior to enrollment:
* A concussive TBI is defined by having at least one of the following after a head trauma (ACRM, 1993) oAny period of loss of consciousness; oAny loss of memory for events immediately before or after the accident; oAny alteration in mental state at the time of the accident (e.g., feeling dazed, disoriented, or confused); and oFocal neurological deficit(s) that may or may not be transient oThe injury must not exceed any of the following (ACRM, 1993):
* Loss of consciousness of approximately 30 minutes or less;
* After 30 minutes an initial GCS score of 13-15; and
* PTA not greater than 24 hours

  * Head trauma resulting in concussive TBI can be due to blast or non-blast mechanisms
  * Head trauma resulting in concussive TBI can have occurred any time in the participant's life: prior to military service, during deployment, in garrison, or after leaving military service
* Have a history of chronic PTH defined as:

  o Headache is reported to have developed (or worsened) after one of the following*:
* The injury to the head;
* Regaining of consciousness following the injury to the head; or
* Discontinuation of medication(s) impairing ability to sense or report headache following the injury to the head
* Not better accounted for by another ICHD-3 diagnosis**

  o The headache persists for >3 months after its onset (ICHD, 2013)
* Have a HIT-6™ score of ≥ 56 to 78 indicative of substantial impact (56-59) or severe impact (60-78) on functioning (Yang, Rendas-Baum, Varon, & Kosinski, 2011)
* Be able to provide written, informed consent in English and follow study-related instructions
* Have ownership of or reliable access to a smartphone with a data plan or internet connecting capabilities
* Be aged ≥ 18 to ≤ 70 years
* Have a history of concussive TBI ≥ 3 months prior to enrollment:
* A concussive TBI is defined by having at least one of the following after a head trauma (ACRM, 1993):

  * Any period of loss of consciousness;
  * Any loss of memory for events immediately before or after the accident;
  * Any alteration in mental state at the time of the accident (e.g., feeling dazed, disoriented, or confused); and
  * Focal neurological deficit(s) that may or may not be transient
  * The injury must not exceed any of the following (ACRM, 1993):
* Loss of consciousness of approximately 30 minutes or less;
* After 30 minutes an initial GCS score of 13-15; and
* PTA not greater than 24 hours

  * Head trauma resulting in concussive TBI can be due to blast or non-blast mechanisms
  * Head trauma resulting in concussive TBI can have occurred any time in the participant's life: prior to military service, during deployment, in garrison, or after leaving military service
* Have a history of chronic PTH defined as:

  o Headache is reported to have developed (or worsened) after one of the following*:
* The injury to the head;
* Regaining of consciousness following the injury to the head; or
* Discontinuation of medication(s) impairing ability to sense or report headache following the injury to the head
* Not better accounted for by another ICHD-3 diagnosis**

  o The headache persists for >3 months after its onset (ICHD, 2013)
* Have a HIT-6™ score of ≥ 56 to 78 indicative of substantial impact (56-59) or severe impact (60-78) on functioning (Yang, Rendas-Baum, Varon, & Kosinski, 2011)
* Be able to provide written, informed consent in English and follow study-related instructions
* Have ownership of or reliable access to a smartphone with a data plan or internet connecting capabilities

Exclusion Criteria:

* They experienced a moderate or severe TBI
* Their secondary headache is better accounted for by the ICHD-3 diagnosis of 8.2 medication-overuse headache; must meet diagnostic criteria for at least 1 medication-overuse headache diagnosis (8.2.1-8.2.8)
* They are currently engaged in psychotherapeutic treatment or have engaged in psychotherapeutic treatment within 8 weeks prior to trial enrollment (for more information regarding recent treatment in potential participants, see section '3.2 Study Procedures,' sub-section 'Baseline Evaluation')
* They report change or discontinuation of headache prophylaxis in the past 4 weeks
* They report active psychotic or bipolar symptoms
* In the opinion of the investigator, they have other considerations that may adversely affect patient safety, participation, or scientific validity of the data being collected (including, but not limited to, active plan or intent for suicide, visual impairment, hand dysfunction or amputation, substantial cognitive impairment, life expectancy of less than 6 months)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
6-Item Headache Impact Test™ (HIT-6™) | 16 weeks
  The HIT-6™ is a brief standardized headache screening tool and questionnaire, derived from the original 54-item Headache Impact Test. It has been found to have good psychometric properties in assessing headache impact among patients in clinical practice and research (Bjorner, Kosinski, & Ware, 2003; Kosinski et al., 2003).

SECONDARY OUTCOMES:
Determine the appropriate sample size for a future full clinical trial based on preliminary estimates of effect size for outcome measures | 12 weeks
  Use of Headache Impact Test and number of headache days per month to compare arms. This data will identify any changes to sample size in future studies.
Post Traumatic Stress Disorder Checklist (DSM-5) | 16 weeks
  The PCL-5 is a self-report questionnaire designed to assess symptoms of PTSD (Blevins, Weathers, Davis, Witte, & Domino, 2015). The PCL-5 takes approximately 5-10 minutes to complete.
Traumatic Brain Injury Quality of Life Scale (TBI-QOL) | 16 weeks
  The TBI-QOL is a self-report questionnaire composed of 22 item banks (Tulsky et al., 2016). It was developed to measure multiple domains of life for patients living with TBI, including physical, mental, cognitive, and social. The TBI-QOL takes approximately 30 minutes to complete.
Patient Health Questionnaire-9 | 16 weeks
  The PHQ-9 is a self-report assessment for depressive symptoms (Kroenke, Spitzer, & Williams, 2001). Each item is scored on a scale of 0 to 3 providing a summary score that ranges from 0 to 27, with higher scores representing more severe depression. On the PHQ-9 a total score <5 is considered minimal depression, and scores of 5 to 9, 10 to 14, 15 to 19, and 20 to 27 are considered mild, moderate, moderately severe, and severe depression, respectively.
Insomnia Severity Index (ISI) | 16 weeks
  The ISI is a self-report questionnaire designed to assess the presence and severity of primary insomnia sleep disorder and is empirically-validated in general and military populations (Bastien et al., 2001; Jenkins et al., 2015; Morin, Belleville, Belanger, & Ivers, 2011).
User Version of the Mobile Application Rating Scale | 12 weeks
  Adapted from the Mobile Application Rating Scale (MARS), the uMARS is a 26-item self-report questionnaire designed to assess the quality, functionality, and aesthetics of a mobile application and its information (Stoyanov, Hides, Kavanagh, & Wilson, 2016). There is an additional open-text question for further comments on the users' opinions of the application. The uMARS takes approximately 15 minutes to complete. This measure will be optional for participants to complete.
Mobile Agnew Relationship Measure | 12 weeks
  The mARM is an adaptation of a valid and reliable assessment of therapeutic alliance in face-to-face therapy (Berry, Salter, Morris, James, & Bucci, 2018). The 25-item questionnaire has been adjusted for use with digital health interventions, specifically for mental health. The mARM takes approximately 5 minutes to complete.
User Program Feedback Questionnaire | 12 weeks
  Brief questionnaire utilizing Likert Scales related to gathering user feedback on personal experience with ease and accessibility of app utilization.

CONTACTS AND LOCATIONS:
Locations (1):
- 100% Remote Recruitment: Center for Neurscience and Regenerative Medicine, Bethesda, Maryland, United States

REFERENCES:
- [Background] Berry K, Salter A, Morris R, James S, Bucci S. Assessing Therapeutic Alliance in the Context of mHealth Interventions for Mental Health Problems: Development of the Mobile Agnew Relationship Measure (mARM) Questionnaire. J Med Internet Res. 2018 Apr 19;20(4):e90. doi: 10.2196/jmir.8252. PMID 29674307
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Wilson H. Development and Validation of the User Version of the Mobile Application Rating Scale (uMARS). JMIR Mhealth Uhealth. 2016 Jun 10;4(2):e72. doi: 10.2196/mhealth.5849. PMID 27287964
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Jenkins MM, Colvonen PJ, Norman SB, Afari N, Allard CB, Drummond SP. Prevalence and Mental Health Correlates of Insomnia in First-Encounter Veterans with and without Military Sexual Trauma. Sleep. 2015 Oct 1;38(10):1547-54. doi: 10.5665/sleep.5044. PMID 26085301
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Tulsky DS, Kisala PA, Victorson D, Carlozzi N, Bushnik T, Sherer M, Choi SW, Heinemann AW, Chiaravalloti N, Sander AM, Englander J, Hanks R, Kolakowsky-Hayner S, Roth E, Gershon R, Rosenthal M, Cella D. TBI-QOL: Development and Calibration of Item Banks to Measure Patient Reported Outcomes Following Traumatic Brain Injury. J Head Trauma Rehabil. 2016 Jan-Feb;31(1):40-51. doi: 10.1097/HTR.0000000000000131. PMID 25931184
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Kosinski M, Bjorner JB, Ware JE Jr, Batenhorst A, Cady RK. The responsiveness of headache impact scales scored using 'classical' and 'modern' psychometric methods: a re-analysis of three clinical trials. Qual Life Res. 2003 Dec;12(8):903-12. doi: 10.1023/a:1026111029376. PMID 14651411
- [Background] Bjorner JB, Kosinski M, Ware JE Jr. Using item response theory to calibrate the Headache Impact Test (HIT) to the metric of traditional headache scales. Qual Life Res. 2003 Dec;12(8):981-1002. doi: 10.1023/a:1026123400242. PMID 14651417